## COMPLUTENSE UNIVERSITY OF MADRID FACULTY OF NURSING, PHYSIOTHERAPY AND PODIATRY



### TITLE:

# CLINICAL TRIAL WITHOUT MEDICATION: PREVENTION OF BODY IMAGE DISORDER FOR NURSING INTERVENTION ON PATIENT AND FAMILY PRIOR TO MAMA AND COLON CANCER SURGERY

## MEMORY TO CHOOSE THE DEGREE OF DOCTOR PRESENTED BY

Natalia Mudarra García

Under the direction of the doctors

Enrique Pacheco Del Cerro Alfonso Meneses Morroy

Madrid, 2018

PREVENTING THE DISORDER OF THE BODY IMAGE IN PATIENT AND FAMILY MEMBERSBY EFFECTIVE HEALTH EDUCATION (NURSING INTERVENTION) PRIOR TO A SURGICAL PROCEDURE OF BREAST AND COLON CANCER.

#### **SUMMARY**

Cancer is one of the most important public health problems worldwide in the 21st century. The National Institute of Neoplastic Diseases emphasizes that cancer of prostate, colon-rectum, lung (in men) and breast and colon-rectum (in women) are among the most common neoplasms.

One of the main treatments to be able to approach this type of tumors, such as breast and colorectal, is surgery. There are different surgical procedures (surgery conservative, mastectomy, ostomy), which, forcefully, have an impact on body image of the individual, sometimes generating extreme and painful situations. These are procedures that lead to biopsychosocial implications and that generate a change in the modus of vivendi.

A better psychological preparation and an effective health education such as nursing intervention of the patient prior to surgery (consisting of providing information about the intervention, giving psychological support in the entire surgical process and reporting on sensations that the patient will experience) will balance the characteristic stressful attribute of surgery and decrease the level of anxiety of the individual.

For the patient to overcome this change in his corporal image, the role of his immediate family is fundamental. Not only because they help to improve the patient's quality of life during his illness, but also because an adequate emotional state of the patient can improve his therapeutic response.

The aim of this study was to assess the body image disorder suffered by patients with breast and colon cancer after surgery. Likewise, the aim was to compare the group of patients and her family members who received an effective health education prior to oncological surgery with patients who did not receive it.

A randomized, non-blinded, controlled clinical trial was conducted. The study consisted of performing a nursing intervention prior to breast and colon surgery to both groups, giving health education divided into four phases: providing information on the disease, showing surgeries and similar experiences, explaining coping methods and reporting on techniques of relaxing.

Statistically significant differences were found between the results of these groups (p <0.001). The study group obtained a lower score on the scale of affectation of the corporal image than the control group.

The most important conclusion is that the fact of performing a care procedure before oncological breast or colon surgery reduces the disorder of the body image in the patient. If this procedure is performed simultaneously on the patient and on an immediate family member, this reduction is even greater.